CLINICAL TRIAL: NCT05384106
Title: AN OPEN-LABEL, ACUTE CLINICAL TRIAL TO ASSESS THE LEVEL OF KETONE PRODUCTION FOLLOWING CONSUMPTION OF AVELA™ (R)-1,3-BUTANEDIOL IN AN ADULT POPULATION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Genomatica Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1129
Record Dates: First submitted 2022-05-12; First posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avela™ (R)-1,3-Butanediol (Experimental): 3 servings of Avela™, with consumption of each serving separated by 30 minutes and each serving providing 11.5 g of (R)-1,3-butanediol [total intake of 34.5 g of (R)-1,3-butanediol].
  Interventions: Dietary Supplement: (R)-1,3-butanediol

INTERVENTIONS:
Dietary Supplement: (R)-1,3-butanediol — Avela™ (R)-1,3-butanediol is intended to induce ketosis in the general adult population. Avela™ (R)-1,3-butanediol is GRAS for use in beverages, bars, and gels
  Other Names: Avela

SUMMARY:
The purpose of the pilot clinical trial described herein is to determine the level of ketone production [measured as β hydroxybutyrate (BHB)] following consumption of (R)-1,3-butanediol in a beverage and to record gastrointestinal (GI) symptomology, as well as any effects on alertness/sleepiness.

DETAILED DESCRIPTION:
Primary:

To evaluate the level of production of BHB following the consumption of 3 servings of Avela™, with consumption of each serving separated by 30 minutes and each serving providing 11.5 g of (R)-1,3-butanediol [total intake of 34.5 g of (R)-1,3-butanediol].

BHB levels will be measured using capillary whole blood from the fingertips using at home Keto-Mojo monitoring system (β-Ketone, as beta-hydroxybutyrate, in fingertip capillary whole blood).

Measurement Range: 0.1 - 8.0 mmol/L Measurement time (min): 0, 30, 60, 90, 120, 180, 240, 300

Secondary:

To evaluate the acute effects of 3 servings of Avela™, with consumption of each serving separated by 30 minutes and each serving providing 11.5 g of (R)-1,3-butanediol [i.e., total intake of 34.5 g (R)-1,3-butanediol] on: GI tolerance.

All subjects will complete the mVAS GI symptoms tool at baseline (0 minutes), and at 30, 60, 90, 120, 180, 240, and 300 minutes.

A validated tool to measure GI tolerability of (R)-1,3-butanediol will be utilized. The mVAS GI symptoms tool is a self-administered questionnaire, which is modeled after the validated "gold standard" measurement tool predominantly used to test clinical gastroenterology scenarios (Bengtsson et al., 2013).

Sleepiness/alertness The SSS (Shahid et al., 2012) is a subjective tool to assess how alert a subject is feeling at specific moments in time. The scale requires respondents to select a rating of 1 to 7, where a "1" indicates the subject is "feeling active, vital, alert, or wide awake" and the highest score of "7" indicates the subject is "no longer fighting sleep, sleep onset soon; having dream-like thoughts" (Hoddes et al., 1973). The scale is validated, correlating r = 0.68 with performance on the Wilkinson tests. All subjects will complete the SSS at baseline (0 minutes) and at 30, 60, 90, 120, 180, 240, and 300 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 to 65 years of age
* BMI 18 to <35.0 kg/m2, inclusive
* Weight ≥ 110 lbs
* Subject is judged to be in good health on the basis of medical history
* Subject is willing to fast for 12 hours prior to study start
* Subject is willing to avoid alcohol and intense physical activity the day prior to and on the day of testing
* Subject is capable of giving informed consent and complying with all study procedures/requirements.

Exclusion Criteria:

* Previous GI disorders (e.g., inflammatory bowel disease, irritable bowel syndrome, history of surgery for weight loss, or gastroparesis)
* Gastroenteritis in the 2 weeks preceding the study
* Diabetes
* Weight <110 lbs
* History of alcohol or drug abuse
* Previous diagnosis of neurological disorders, depression, or mental illness with psychosis
* Unexplained alarm features (i.e., unintentional weight loss >10% body weight in the last 3 months, fevers, or blood in stools)
* Use of an antibiotic or any medication impacting gut transit during the 2 weeks before the study
* Constipation or diarrhea (defined as, on average, less than 3 stools per week or more than 3 stools per day, respectively)
* Allergy to tree nuts
* Women who are pregnant or breastfeeding
* Persons with medical conditions affecting the pancreas, liver, thyroid, or gall bladder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-25 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the level of production of BHB measure of blood ketones levels (i.e., blood BHB levels) | 0, 30, 60, 90, 120, 180, 240, and 300 minutes
  β-Ketone, as beta-hydroxybutyrate, in fingertip capillary whole blood, Measurement Range: 0.1 - 8.0 mmol/L

SECONDARY OUTCOMES:
To assess GI symptomology | 0, 30, 60, 90, 120, 180, 240, and 300 minutes
  Modified visual analogue scale (mVAS) GI symptoms tool
To assess Sleepiness/alertness | 0, 30, 60, 90, 120, 180, 240, and 300 minutes
  Stanford Sleepiness Scale (SSS)

CONTACTS AND LOCATIONS:
Locations (1):
- Moniker Commons, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT05384106/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT05384106/ICF_001.pdf